CLINICAL TRIAL: NCT06367504
Title: A Randomized, Double-blind, Placebo-controlled, Pilot Clinical Study to Assess the Effect of Doctor's Biome Medical Food (DBMF) in Individuals With Clostridium Difficile Infection (CDI)
Brief Title: A Study to Assess the Effect of Doctor's Biome Medical Food in Individuals With Clostridium Difficile Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DB/230904/DBMF/CDI
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-03

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doctor's Biome Medical Food (DBMF) (Active Comparator): Once a day daily 30 minutes before lunch
  Interventions: Dietary Supplement: DBMF
- Placebo (Placebo Comparator): Once a day daily 30 minutes before lunch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DBMF — Once a day daily 30 minutes before lunch
  Arms: Doctor's Biome Medical Food (DBMF)
Dietary Supplement: Placebo — Once a day daily 30 minutes before lunch
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, pilot clinical study to assess the effect of Doctor's Biome Medical Food (DBMF) in individuals with Clostridium difficile infection (CDI)

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of 30 - 75 years of age.
2. A qualifying episode of CDI as defined by:

   1. ≥ 3 abnormal stools as assessed by BSFS score of 6 & 7 in the last 24 hours.
   2. A positive C. difficile stool toxin assay as assessed by C. difficile toxins A & B - CARD*.
   3. The requirement of CDI Standard of Care (SOC) antibiotic therapy (as per PI's discretion). 3) Individuals willing to give voluntary, written informed consent to participate in the study.

4) Individuals without/with antibiotic-associated diarrhea (indicated by use of antibiotics any time in last one week) will also be considered for the testing of C. difficile toxins

Exclusion Criteria:

1. History or presence of terminal/end-stage renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders (which might confound the interpretation of the study results, or put the individual at undue risk).
2. History of peptic ulcer.
3. History of abdominal surgery within the previous 3 months.
4. Presence of colostomy, gastric-tube, or naso-gastric-tube.
5. Individuals requiring any gastrointestinal surgery planned during the next 3 months.
6. HIV, AIDS, primarily immunodeficiency, cancer
7. Individuals with a very recent (< 1 year) solid organ or bone marrow transplant.
8. Individuals requiring blood transfusion or renal dialysis planned during the next 3 months.
9. Unwilling to abstain using kombucha, sauerkraut, pickles and kimchi
10. Individuals with the following food intolerance - gluten, lactose, and/or histamine.
11. Heavy alcohol drinkers are defined as follows: For men, consuming more than 4 drinks on any day or more than 14 drinks/week. For women, consuming more than 3 drinks on any day or more than 7 drinks/week.
12. Smokers.
13. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
14. Individuals who have participated in another clinical study(ies) with an investigational product within 90 days before screening, or who plan to participate in another study during the study period.
15. Use of any supplements (may include probiotics, post-biotics, herbal supplements, synbiotics, enzyme supplementation the last 30 days.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of Investigational product on the duration of Clostridium difficile diarrhea in comparison to placebo. | Day 0, day 28 and day 56
  The Clostridium difficile Toxin A+B Card is a non-invasive, rapid immunochromatographic test for detecting toxins A and B in stool samples for making a presumptive diagnosis of Clostridium difficile infection.

SECONDARY OUTCOMES:
To assess the impact of the Investigational product on Number of CDI diarrhea episodes presence of Clostridium difficile in stool samples as assessed by C. difficile toxins A & B - CARD. | day 28 and day 56
  The Clostridium difficile Toxin A+B Card is a non-invasive, rapid immunochromatographic test for detecting toxins A and B in stool samples for making a presumptive diagnosis of Clostridium difficile infection.
To assess the impact of the Investigational product on Change in the frequency of watery stools from Bristol Stool Form Scale (BSFS) score type 7 as compared to placebo. | throughout the study during diarrhea episodes upto day 56
  Bristol Stool Form Scale (BSFS), a simple and inexpensive tool that categorizes the stool into one of seven stool types ranging from type 1 (hard lumps) to type 7 (watery diarrhea). Stool consistency (diarrhea) serves as a surrogate marker for a C. difficile infection
To assess the impact of the Investigational product on Number of non-CDI diarrhea episodes as compared to placebo | day 28 and day 56
  Participants with frequency of ≥ 3 abnormal stools as assessed by BSFS stool type 6 &/or 7 for 1 day will be analyzed for the presence of CDI using the CARD test.
To assess the impact of the Investigational product on Number of SOC medication consumed (antibiotics therapy) throughout the intervention period as compared to placebo. | throughout the study during diarrhea episodes upto day 56
  Antibiotics induce adverse changes in gut microbiota, leading to a reduction in the absorption of short-chain fatty acids, resulting in osmotic, or watery, diarrhea
To assess the impact of the Investigational product on Average number of days of consumption of SOC (antibiotics therapy) as compared to placebo. | throughout the study during diarrhea episodes upto day 56
  Antibiotics induce adverse changes in gut microbiota, leading to a reduction in the absorption of short-chain fatty acids, resulting in osmotic, or watery, diarrhea

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - AIMS Hospital, Dombivali, Maharashtra
  - Stress Test Clinic, Mumbai, Maharashtra
  - Nobel Hospital, Pune, Maharashtra
  - Gleneagles Hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No